CLINICAL TRIAL: NCT03298971
Title: The Impact of Cancer and Treatment-related Effects on the Physical and Psychosocial Well-being and Quality of Life Among Hong Kong Chinese Survivors of Childhood Osteosarcoma: An Exploratory Study
Brief Title: The Impact of Cancer on the Physical and Psychosocial Well-being Among Childhood Osteosarcoma Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 17-331
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-11

CONDITIONS: Childhood Osteosarcoma
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors of Childhood Osteosarcoma: Survivors of Childhood Osteosarcoma were invited to fill in a set of questionnaires.
  Interventions: Other: Questionnaires
- Healthy Subjects: Healthy Subjects were invited to fill in a set of questionnaires.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants were asked to respond to the questionnaires including Hong Kong Chinese Version World Health Organization quality of life measure, abbreviated version (WHOQOL-BREF (HK)), the Chinese version of The Center for Epidemiological Studies - Depression Scale (CES-D), the Chinese version of Rosenberg self-esteem scale, and the Chinese version of the Herth Hope Index (HHI).

SUMMARY:
The aim of the study is to examine the impact of cancer and treatment-related effects on the physical and psychosocial well-being and quality of life among Hong Kong Chinese survivors of childhood osteosarcoma.

DETAILED DESCRIPTION:
Osteosarcoma is the most common primary malignant bone tumor in children and adolescents. The 5-year overall survival rates of childhood osteosarcoma survivors have been increasing substantially with a percentage approaching to 70%. Regrettably, the improved survival rates may lead to long-term sequelae related to disease and treatments that can negatively affect survivors' physical and psychological well-being. Despite numerous studies have examined the impact of cancer and treatment-related late effects on the physical and psychological aspects of osteosarcoma survivors in the foreign countries, it has not been studied specifically in Hong Kong Chinese population. Problems arise when there is a difference in perception and recognition of psychological problems and emotional well-being between Western and Chinese culture. Moreover, the difference in coping strategies between Chinese and Western children also affects how they react and cope with the devastating effect from cancer and its treatments. Due to the cultural and belief differences, the findings from those studies in the foreign counties may not be applicable and transferable in Hong Kong context. There is thus an imperative need to investigate the impact of cancer and treatment-related effects on the physical and psychosocial well-being and quality of life among Hong Kong Chinese survivors of childhood osteosarcoma in order to raise awareness of the holistic wellness of osteosarcoma survivors.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese under the age of 30 years at the time of study participation;
* Diagnosed with osteosarcoma under the age of 19 years;
* Completed the entire course of treatment at least 5 years;
* Able to speak fluent Cantonese and read Chinese.

Exclusion Criteria:

* Survivors with secondary malignancy, organic cause psychosis, cognitive or learning problems, or under active cancer treatment

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hong Kong Chinese under the age of 30 years who completed the entire course of treatment at least 5 years and were diagnosed with osteosarcoma under the age of 19 years.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Levels of quality of life at baseline | baseline
  The quality of life of the participants will be measured by the Hong Kong Chinese Version World Health Organization quality of life measure, abbreviated version (WHOQOL-BREF (HK)). It consists of 28 items with a five-point response Likert scale. There are two questions to access the overall perception of quality of life and health respectively. The remaining 26 items were designed to assess the perception of quality of life in four particular domains including physical health, psychological well-being, social relationships and environments. Higher scores represent higher levels of QoL. Participants will be asked to respond to the Hong Kong Chinese Version World Health Organization quality of life measure, abbreviated version (WHOQOL-BREF (HK)) at baseline.

SECONDARY OUTCOMES:
Levels of self-esteem at baseline | baseline
  The self-esteem of the participants will be measured by the Chinese version of the Rosenberg Self-esteem Scale (RSES). RSES consists of 10 items with a four-point response Likert scale ranging from 1 (strongly agree) to 4 (strongly disagree) and the total scores is ranging from 10 to 40. Higher scores represent higher levels of self-esteem. Participants will be asked to respond to the Chinese version of the Rosenberg Self-esteem Scale (RSES) at baseline.
Number of depressive symptoms at baseline | baseline
  The number of depressive symptoms of the participants will be measured by the Center for Epidemiological Studies - Depression Scale (CES-D). It is able to assess the numbers of depressive symptoms due to the experience of past week. The scale consists of 20 items with four-point Likert scale for patients to response and the total score is ranging from 0 to 60. Higher scores represent greater numbers of depressive symptoms while lower scores represent fewer numbers of depressive symptoms. Participants will be asked to respond to the Center for Epidemiological Studies - Depression Scale (CES-D) at baseline.
Level of sense of hope at baseline | baseline
  The sense of hope of the participants will be measured by the Chinese version of Herth Hope Index (HHI). It is a 12-item psychometric scale to measure the sense of hope. Each item contains four-point scale ("strong disagree" = "1", "disagree" = "2", "agree" = "3", "strong agree" = "4"). The total score of the 12 items ranging from 12 to 48 and higher scores imply increasing hopefulness. Participants will be asked to respond to the Chinese version of the Herth Hope Index (HHI) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No